CLINICAL TRIAL: NCT03032978
Title: Clinical and Microbiological Evaluation of Calcium Silicate Versus Calcium Hydroxide in Two-step Indirect Pulp Treatment: Randomized Clinical Trial
Brief Title: Calcium Silicate Versus Calcium Hydroxide in Two-step Indirect Pulp Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ehsan hossam, Assistant lecturer conservative dentistry - Ahram canadian university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2017-01-06
Record Dates: First submitted 2017-01-14; First posted 2017-01-26 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Deep Caries
MeSH Terms: interventions — Calcium Hydroxide; Dycal; calcium silicate; TheraCal

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Calcium silicate (Experimental): intervention
  Interventions: Other: Calcium silicate
- Calcium Hydroxide (Active Comparator): Comparator
  Interventions: Other: Calcium hydroxide

INTERVENTIONS:
Other: Calcium hydroxide — Pulp capping material
  Other Names: Dycal
  Arms: Calcium Hydroxide
Other: Calcium silicate — Pulp capping material
  Other Names: Theracal
  Arms: Calcium silicate

SUMMARY:
Clinical and microbiological evaluation of Calcium silicate versus Calcium hydroxide in two-step indirect pulp treatment: Randomized clinical trial

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years.
* Males or females.
* Co-operative patients approving to participate in the trial.

Exclusion Criteria:

* Patients younger than 19 years old or older than 50 years old.
* Disabilities.
* Systemic diseases or severe medically compromised.
* Lack of compliance.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Pain: VAS | 6 month
  post operative pain after 6 month from material application will be measured by visual analogue scale (VAS)with score from 0 to 10 in which 0 means no pain and 10 means the worst pain

CONTACTS AND LOCATIONS:
Locations (1):
- Ehsan Hossam, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided